CLINICAL TRIAL: NCT04470544
Title: RECOVER: Phase 2 Randomized, Double-Blind Trial TREating Hospitalized Patients With COVID-19 With Camostat MesilatE, a TMPRSS2 Inhibitor
Brief Title: Camostat Mesilate Treating Patients With Hospitalized Patients With COVID-19
Acronym: RECOVER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alan Bryce (Other)
Responsible Party: Sponsor-Investigator, Alan Bryce, Principal Investigator, Academic and Community Cancer Research United
Organization: Academic and Community Cancer Research United (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAM20CV
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-02

CONDITIONS: Severe Acute Respiratory Syndrome
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — camostat; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo + Standard of Care (Placebo Comparator): Standard of Care will be defined by the investigators in collaboration with the sponsor on the basis of the best available evidence at the time of study initiation with placebo.
  Interventions: Other: Standard of Care
- Camostat + Standard of Care (Experimental): Patient will receive SOC tablets and Camostat mesilate 200 mg four times a day after each meal with Standard of Care treatment.
  Interventions: Drug: Camostat Mesilate

INTERVENTIONS:
Drug: Camostat Mesilate — Given PO
  Other Names: Foipan
  Arms: Camostat + Standard of Care
Other: Standard of Care — At Investigator discretion
  Arms: Placebo + Standard of Care

SUMMARY:
To determine if the reduction in TMPRSS2 activity via direct inhibition with Camostat mesilate combined with standard of care (SOC) treatment will increase the proportion of patients alive and free from respiratory failure at Day 28 in SARS-CoV-2 as compared to SOC treatment with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed SARS-CoV-2 infection
* Admitted to hospital for management of SARS-CoV-2
* Age ≥18
* Subject or legal representative able to give informed consent
* Ability to take all study drugs
* Respiratory status of 3 or greater on the WHO ordinal scale
* ALT or AST ≤5 x ULN
* Creatinine clearance ≥50 mL/min using the Cockroft-Gault formula
* Willingness to provide mandatory specimens for correlative research and banking

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Known hypersensitivity to the study drug, the metabolites or formulation excipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan H Bryce, M.D., Principal Investigator — Academic and Community Cancer Research United
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Tucson Medical Center, Tucson, Arizona

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo + Standard of Care | Camostat + Standard of Care
Started | 50 | 50
Completed | 46 | 44
Not Completed | 4 | 6
Not completed — Withdrawal by Subject | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Standard of Care will be defined by the investigators in collaboration with the sponsor on the basis of the best available evidence at the time of study initiation with placebo.
- Camostat: Patient will receive SOC tablets and Camostat mesilate 200 mg four times a day after each meal with Standard of Care treatment.
- Total: Total of all reporting groups
Arm/Group | Placebo | Camostat | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (15.7) | 57.1 (18.4) | 57.7 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 34 | 32 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 15
  Not Hispanic or Latino | 41 | 39 | 80
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 40 | 41 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Alive and Free From Respiratory Failure
Description: To determine if the reduction in TMPRSS2 activity via direct inhibition with Camostat mesilate combined with standard of care (SOC) treatment will change the proportion of patients alive and free from respiratory failure at Day 28 in SARS-CoV-2 as compared to SOC treatment with placebo.
Time Frame: 28 Days
Population: All patients that submitted day 28 outcome data
Measure: Number; unit: Proportion of patients
Arm/Group | Placebo | Camostat
Number analyzed (Participants) | 46 | 43
Proportion of patients | .891 | .884

2. Secondary Outcome: Proportion of Patients Alive and Free of Ventilator Use or ECMO
Description: To determine if reduction in TMPRSS2 activity via direct inhibition with Camostat mesilate combined with SOC treatment will change the proportion of patients alive and free of ventilator use or ECMO at Day 28 as compared to SOC treatment combined with placebo.
Time Frame: 28 Days
Population: All patients that submitted day 28 outcome data
Measure: Number; unit: Proportion of patients
Arm/Group | Placebo | Camostat
Number analyzed (Participants) | 46 | 43
Proportion of patients | .891 | .883

3. Secondary Outcome: Mortality Rate
Description: To determine if the combination of Camostat mesilate combined with SOC treatment will result in a changed mortality rate at 28 days as compared to SOC treatment combined with placebo.
Time Frame: 28 Days
Population: All patients that submitted day 28 outcome data
Measure: Number; unit: proportion of participants
Arm/Group | Placebo | Camostat
Number analyzed (Participants) | 46 | 43
proportion of participants | .061 | .070

4. Secondary Outcome: Clinical Change
Description: Clinical change will be defined as a 2 or more point decease on the WHO ordinal scale. The WHO ordinal scale ranges from 0, the best status, to 8, death. Time to clinical improvement will be calculated as the number of days from study entry until the earliest date of clinical change.
Time Frame: 28 Days
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Camostat
Number analyzed (Participants) | 46 | 44
Days | 4 [3 to 5] | 4 [3 to 5]

5. Secondary Outcome: Adverse Event Grade 3 Plus Rate
Description: Analyses for safety will include all participants who are randomized and received at least 1 dose of study treatment. Participants will be grouped according to the treatment to which they were randomized.
Time Frame: 28 days
Population: All treated patients that were evaluated for adverse events.
Measure: Number; unit: proportion of participants
Arm/Group | Placebo | Camostat
Number analyzed (Participants) | 46 | 44
proportion of participants | .17 | .20

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | Placebo | Camostat
All-Cause Mortality (participants affected / at risk) | 4/50 | 3/50
Serious Adverse Events (participants affected / at risk) | 4/50 | 2/50
Other Adverse Events (participants affected / at risk) | 16/50 | 21/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=50) | Camostat (N=50)
Death NOS (General disorders) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=50) | Camostat (N=50)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 1 (1) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Shingles (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Weight gain (Investigations) | 0 (0) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT04470544/Prot_SAP_000.pdf